CLINICAL TRIAL: NCT05748028
Title: Pain and Autonomic Symptoms in Parkinson's Disease and Atypical Parkinsonisms: Identification of Predictive Patterns of Rehabilitation Outcome and Evaluation of the Impact on Quality of Life
Brief Title: Pain and Autonomic Symptoms in Parkinson's Disease and Atypical Parkinsonisms
Status: Recruiting | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Other Study IDs: SBLAB1/19
Record Dates: First submitted 2023-01-26; First posted 2023-02-28 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease; Multiple System Atrophy
Keywords: pain; autonomic symptoms; rehabilitation
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; Pain | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson Disease: Patients affected by Parkinson's disease admitted for rehabilitation in Maugeri Clinical Scientific Institutes
  Interventions: Other: Rehabilitation; Other: Administration of Clinical scales
- Multiple System Atrophy: Patients affected by Multiple System Atrophy admitted for rehabilitation in Maugeri Clinical Scientific Institutes
  Interventions: Other: Rehabilitation; Other: Administration of Clinical scales

INTERVENTIONS:
Other: Rehabilitation — All patients included in the study will undergo a basic evaluation with a neurological examination, a rehabilitation program to improve strength, coordination, balance, endurance, and the ability to perform activities of daily life.
Other: Administration of Clinical scales — All patients included in the study will be evaluated by clinical scales assessing the disease stage, clinical severity, freezing, motor and non-motor impairment, cognitive impairment, depression, quality of life, autonomic dysfunction, pain.

SUMMARY:
The goal of this observational study is to learn about the impact of the different types of pain and of the domains involved in the autonomic disorders of inpatients and outpatients diagnosed with Parkinson disease (PD) and multiple system atrophy (MSA) admitted to Istituti Clinici Scientifici Maugeri Centers.

The main aims are:

Evaluate the prevalence of pain and characterize it in Parkinson's disease and atypical parkinsonisms (MSA) Evaluate the effect of rehabilitation on pain and autonomic symptoms Evaluate the prevalence of autonomic symptoms in Parkinson's disease and atypical parkinsonisms (MSA) Assess the impact of pain and autonomic symptoms on quality of life. Participants will perform neurological examination, rehabilitation program and clinical scales.

Researchers will compare the two groups of patients (PD and MSA) and the effect of the rehabilitation on pain, autonomic symptoms and quality of life.

DETAILED DESCRIPTION:
2% of the population over 65 is affected by Parkinson's disease (PD) or parkinsonism. This represents a significant burden on the health service in countries where the elderly represent 1/5 of the general population. In recent years there has been increased attention on the presence of non-motor disorders in PD patients. Among these, pain and autonomic symptoms are more frequently present and contribute to the worsening of disability and quality of life of the affected patient.

How much the presence of pain and autonomic symptoms can affect the rehabilitation outcome and how much the rehabilitation treatment itself can improve the painful or autonomic symptomatology is not known, but rehabilitation has an important role in the management of diseases where there are no real treatments capable of cure or slow down the neurodegenerative process.

In the Maugeri Clinical Scientific Institutes, patients with Parkinson's disease or parkinsonism are hospitalized or followed as outpatients and a personalized rehabilitation setting is ideal for being able to evaluate the patient in a sufficiently wide time frame to be able to appreciate significant changes in clinical parameters.

The greater knowledge of the impact of the different types of pain and of the domains involved in the autonomic dysfunction will help the clinician to better manage the patient's disability and will contribute to the definition of specific rehabilitation strategies aimed to improve the patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's Disease or Multiple System Atrophy according to current international criteria (Gilman S et al, 2008; Postuma RB et al. 2015).
* Mini-Mental State Examination score at least 10

Exclusion Criteria:

* vascular or pharmacological parkinsonism
* diabetes mellitus
* hepatic or renal dysmetabolism,
* hypothyroidism or hyperthyroidism
* assumption of potentially neurotoxic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled from the population of inpatient and outpatient admitted for rehabilitation to ICS Maugeri SpA institutes.
Sampling Method: Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2019-06-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence and Characterization of Pain | At the recruitment
  Evaluate the prevalence of pain and characterize it in Parkinson's disease and atypical parkinsonisms through KING'S PAIN score
Prevalence and Characterization of Pain | At the end of the rehabilitation program, an average of 30 days
  Evaluate the prevalence of pain and characterize it in Parkinson's disease and atypical parkinsonisms through KING'S PAIN score

SECONDARY OUTCOMES:
Autonomic symptoms | At the recruitment
  Evaluate the prevalence of autonomic symptoms in Parkinson's disease and atypical parkinsonisms through the score of SCOPA-AUT questionnaire
Autonomic symptoms | At the end of the rehabilitation program, an average of 30 days
  Evaluate the prevalence of autonomic symptoms in Parkinson's disease and atypical parkinsonisms through the score of SCOPA-AUT questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Maria Nolano, MD, PhD, Principal Investigator — Isituti Clinici Scientifici Maugeri SpA SB - IRCCS of Telese Terme
Locations (9):
- Italy (9):
  - ICS Maugeri - IRCCS of Telese Terme, Telese Terme, Benevento
  - ICS Maugeri - Lumezzane, Lumezzane, Brescia
  - ICS Maugeri - Castelgoffredo, Castel Goffredo, Mantova
  - ICS Maugeri - Mistretta, Mistretta, Messina
  - ICS Maugeri - Veruno, Veruno, Novara
  - ICS Maugeri - Montescano, Montescano, Pavia
  - ICS Maugeri - Milano, Milan
  - ICS Maugeri - Pavia Boezio, Pavia
  - ICS Maugeri - Pavia, Pavia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bakkers M, Faber CG, Hoeijmakers JG, Lauria G, Merkies IS. Small fibers, large impact: quality of life in small-fiber neuropathy. Muscle Nerve. 2014 Mar;49(3):329-36. doi: 10.1002/mus.23910. Epub 2013 Jun 28. PMID 23716362
- [Background] Quittenbaum BH, Grahn B. Quality of life and pain in Parkinson's disease: a controlled cross-sectional study. Parkinsonism Relat Disord. 2004 Mar;10(3):129-36. doi: 10.1016/j.parkreldis.2003.12.001. PMID 15036166
- [Background] Valkovic P, Minar M, Singliarova H, Harsany J, Hanakova M, Martinkova J, Benetin J. Pain in Parkinson's Disease: A Cross-Sectional Study of Its Prevalence, Types, and Relationship to Depression and Quality of Life. PLoS One. 2015 Aug 26;10(8):e0136541. doi: 10.1371/journal.pone.0136541. eCollection 2015. PMID 26309254
- [Background] Nolano M, Provitera V, Estraneo A, Selim MM, Caporaso G, Stancanelli A, Saltalamacchia AM, Lanzillo B, Santoro L. Sensory deficit in Parkinson's disease: evidence of a cutaneous denervation. Brain. 2008 Jul;131(Pt 7):1903-11. doi: 10.1093/brain/awn102. Epub 2008 May 31. PMID 18515869
- [Background] Asahina M, Vichayanrat E, Low DA, Iodice V, Mathias CJ. Autonomic dysfunction in parkinsonian disorders: assessment and pathophysiology. J Neurol Neurosurg Psychiatry. 2013 Jun;84(6):674-80. doi: 10.1136/jnnp-2012-303135. Epub 2012 Sep 1. PMID 22942216
- [Background] Linder J, Stenlund H, Forsgren L. Incidence of Parkinson's disease and parkinsonism in northern Sweden: a population-based study. Mov Disord. 2010 Feb 15;25(3):341-8. doi: 10.1002/mds.22987. PMID 20108376
- [Background] Chaudhuri KR, Rizos A, Trenkwalder C, Rascol O, Pal S, Martino D, Carroll C, Paviour D, Falup-Pecurariu C, Kessel B, Silverdale M, Todorova A, Sauerbier A, Odin P, Antonini A, Martinez-Martin P; EUROPAR and the IPMDS Non Motor PD Study Group. King's Parkinson's disease pain scale, the first scale for pain in PD: An international validation. Mov Disord. 2015 Oct;30(12):1623-31. doi: 10.1002/mds.26270. Epub 2015 Jun 11. PMID 26096067
- [Background] Rodriguez-Violante M, Alvarado-Bolanos A, Cervantes-Arriaga A, Martinez-Martin P, Rizos A, Chaudhuri KR. Clinical Determinants of Parkinson's Disease-associated Pain Using the King's Parkinson's Disease Pain Scale. Mov Disord Clin Pract. 2017 Feb 6;4(4):545-551. doi: 10.1002/mdc3.12469. eCollection 2017 Jul-Aug. PMID 30363423
- [Background] Postuma RB, Berg D, Stern M, Poewe W, Olanow CW, Oertel W, Obeso J, Marek K, Litvan I, Lang AE, Halliday G, Goetz CG, Gasser T, Dubois B, Chan P, Bloem BR, Adler CH, Deuschl G. MDS clinical diagnostic criteria for Parkinson's disease. Mov Disord. 2015 Oct;30(12):1591-601. doi: 10.1002/mds.26424. PMID 26474316
- [Background] Gilman S, Wenning GK, Low PA, Brooks DJ, Mathias CJ, Trojanowski JQ, Wood NW, Colosimo C, Durr A, Fowler CJ, Kaufmann H, Klockgether T, Lees A, Poewe W, Quinn N, Revesz T, Robertson D, Sandroni P, Seppi K, Vidailhet M. Second consensus statement on the diagnosis of multiple system atrophy. Neurology. 2008 Aug 26;71(9):670-6. doi: 10.1212/01.wnl.0000324625.00404.15. PMID 18725592